CLINICAL TRIAL: NCT00607659
Title: Immunopathogenesis of Chlamydia Trachomatis Infection
Brief Title: Immunopathogenesis of Chlamydia
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB #99416; Chaos # 1634-2; NIH 5 R01 AI051417-04
Record Dates: First submitted 2008-01-08; First posted 2008-02-06 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: CHLAMYDIA INFECTIONS
Keywords: Chlamydia; Chlamydia trachomatis; Adolescent Health; Female Health; Sexually Transmitted Infections; Infertility; Pelvic Inflammatory Disease
MeSH Terms: conditions — Chlamydia Infections; Sexually Transmitted Diseases; Infertility; Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endocervical or vaginal swabs, rectal swabs, blood (whole and serum),urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chlamydia Positive: Adolescent females, 11-21 years old, evaluated for pelvic examinations or STI screening will be asked to participate in this study. Participants are being asked to give us permission to collect:additional cervical or vaginal swabs, rectal swabs, blood draws where three tablespoons of blood, a urine pregnancy test, and a comprehensive health history. You may be asked to provide a urine specimen at the initial visit instead of having a cervical swab. The study team will obtain a cervical swab when you come back for your follow-up appointments. If your culture is positive for Chlamydia, you will be asked attend 3 additional follow-up appointments after 3 months, 6 months, 1 year, 2 years, and 3 years .
  Interventions: Other: No intervention, only observational
- Control/Chlamydia Negative: Some participants with negative cultures will be included in this study as a control group. The same specimens, exams and blood draws will apply for those subjects with visits at 3 months, 6 months, 1 year, 2 years, and 3 years
  Interventions: Other: No intervention, only observational

INTERVENTIONS:
Other: No intervention, only observational — No intervention, only observational

SUMMARY:
Sexually transmitted Chlamydia trachomatis infections are a widespread public health concern due to their prevalence and potentially devastating reproductive consequences, including pelvic inflammatory disease, infertility, and ectopic pregnancy. The goal of this study is to evaluate the risk factors for adverse outcomes following genital tract infection with Chlamydia trachomatis and to evaluate whether or not the presence of C. trachomatis in the rectum act as a reservoir for infection.

DETAILED DESCRIPTION:
Sexually transmitted Chlamydia trachomatis infections are a widespread public health concern due to their prevalence and potentially devastating reproductive consequences, including pelvic inflammatory disease, infertility, and ectopic pregnancy. The goal of this study is to evaluate the risk factors for adverse outcomes following genital tract infection with Chlamydia trachomatis and to evaluate whether or not the presence of C. trachomatis in the rectum act as a reservoir for infection. Our target population will be adolescent females age 11-21 evaluated at the ACH Adolescent Center who are undergoing pelvic examinations or urine screening for sexually transmitted infections (STIs). Laboratory specimens obtained will include cervical and rectal swabs, urine and blood specimens, as well as, chart review and comprehensive subject interviews in the initial data collection with follow-up evaluations at 3, 6, 12, 24 and 36 months for qualifying subjects

ELIGIBILITY:
Inclusion Criteria:

* Female
* 11 to 21 years of age at the time of enrollment
* Positive for Chlamydia infections by urine or cervical PCR
* 5th Chlamydia-negative subject who fits all other inclusion criteria
* Negative pregnancy test
* Written informed consent provided
* Signed a HIPAA authorization form
* Willingness to comply with all the requirements of the protocol

Exclusion Criteria:

* Positive pregnancy test
* Negative for Chlamydia, unless 5th negative subject to be in the control group
* Any condition that in the opinion of the investigator would interfere with the ability of the potential subject to complete the study or would result in significant risk to the subject

Ages: 11 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent females between 11 and 21 years of age undergoing pelvic examinations or screening for STIs at the Arkansas Children's Hospital Adolescent Center will be eligible for recruitment
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the environmental and behavioral risk factors that predispose toward adverse reproductive outcomes following C. trachomatis genital tract infection in a high risk adolescent population | enrollment,3,6,12,24,36 months

SECONDARY OUTCOMES:
Determine the prevalence of rectal C. trachomatis colonization in this high risk population and its contribution to recurrent and persistent infection and adverse reproductive outcomes such as infertility and ectopic pregnancy | enrollment,3,6,12,24,36 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Scurlock, M.D., Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Igietseme JU, Portis JL, Perry LL. Inflammation and clearance of Chlamydia trachomatis in enteric and nonenteric mucosae. Infect Immun. 2001 Mar;69(3):1832-40. doi: 10.1128/IAI.69.3.1832-1840.2001. PMID 11179361
- [Background] Cotter TW, Ramsey KH, Miranpuri GS, Poulsen CE, Byrne GI. Dissemination of Chlamydia trachomatis chronic genital tract infection in gamma interferon gene knockout mice. Infect Immun. 1997 Jun;65(6):2145-52. doi: 10.1128/iai.65.6.2145-2152.1997. PMID 9169744
- [Background] Jones RB, Rabinovitch RA, Katz BP, Batteiger BE, Quinn TS, Terho P, Lapworth MA. Chlamydia trachomatis in the pharynx and rectum of heterosexual patients at risk for genital infection. Ann Intern Med. 1985 Jun;102(6):757-62. doi: 10.7326/0003-4819-102-6-757. PMID 3888022
- [Background] Dean D, Suchland RJ, Stamm WE. Evidence for long-term cervical persistence of Chlamydia trachomatis by omp1 genotyping. J Infect Dis. 2000 Sep;182(3):909-16. doi: 10.1086/315778. Epub 2000 Aug 17. PMID 10950788
- [Background] Centers for Disease Control and Prevention (CDC). Chlamydia trachomatis genital infections--United States, 1995. MMWR Morb Mortal Wkly Rep. 1997 Mar 7;46(9):193-8. PMID 9072679
- [Background] Darville T. Chlamydia trachomatis infections in neonates and young children. Semin Pediatr Infect Dis. 2005 Oct;16(4):235-44. doi: 10.1053/j.spid.2005.06.004. PMID 16210104
- See also: Arkansas Children's Hospital Main Page — http://www.archildrens.org